CLINICAL TRIAL: NCT05859009
Title: EUS-guided Therapy vs Non-selective Beta Blocker for the Primary Prophylaxis of Gastric Varices Bleed: a Randomized Controlled Trial
Brief Title: Primary Prevention of Gastric Varices Bleed
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No study oversight due to changes in study personnel.
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 23-066
Record Dates: First submitted 2023-03-27; First posted 2023-05-15 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Gastric Varices Bleeding; Endoscopic Ultrasound
MeSH Terms: interventions — p80-coilin; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EUS-Guided Therapy of glue and coil + Non-selective Beta Blockers (Propanolol) (Active Comparator): Participants in this arm will receive a daily oral dose of a non-selective beta blocker (Propanolol) and undergo EUS-guided therapy of glue and coil as described in Arms 1 and 2. Participants will be monitored for side effects, complications, and efficacy of both the medication and the procedure.
  Interventions: Procedure: EUS-Guided Therapy of Glue and Coil; Drug: Non-Selective Beta Blockers (Propanolol)
- EUS-Guided Therapy of Glue and Coil (Active Comparator): Participants in this arm will undergo endoscopic ultrasound (EUS) to identify and target gastric varices. Under EUS guidance, a combination of glue and coil will be used to occlude the gastric varices. Participants will be monitored for complications and efficacy of the procedure
  Interventions: Procedure: EUS-Guided Therapy of Glue and Coil
- Non-Selective Beta Blockers (Propanolol) (Active Comparator): Participants in this arm will receive a daily oral dose of a non-selective beta blocker (such as propranolol) for the duration of the study. Participants will be monitored for side effects and efficacy of the medication.
  Interventions: Drug: Non-Selective Beta Blockers (Propanolol)

INTERVENTIONS:
Procedure: EUS-Guided Therapy of Glue and Coil — This clinical trial aims to evaluate the effectiveness and safety of endoscopic ultrasound (EUS)-guided therapy of glue and coil in the management of gastrointestinal bleeding due to varices. The procedure involves the insertion of a catheter through an endoscope to deliver glue and/or coils to the bleeding site, under EUS guidance. Patients who meet the inclusion criteria will undergo EUS-guided therapy of glue and coil, followed by follow-up assessments to evaluate the outcomes of the procedure, including bleeding recurrence and adverse events.
  Arms: EUS-Guided Therapy of Glue and Coil; EUS-Guided Therapy of glue and coil + Non-selective Beta Blockers (Propanolol)
Drug: Non-Selective Beta Blockers (Propanolol) — Participants in this arm will receive a daily oral dose of a non-selective beta blocker (such as propranolol) for the duration of the study. Participants will be monitored for side effects and efficacy of the medication.
  Other Names: Propanolol
  Arms: EUS-Guided Therapy of glue and coil + Non-selective Beta Blockers (Propanolol); Non-Selective Beta Blockers (Propanolol)

SUMMARY:
Primary prophylaxis of gastric varices is an important area of research, as gastric varices are a common complication of cirrhosis of the liver. Cirrhosis is a condition in which the liver becomes scarred and loses its ability to function properly, and it is a leading cause of morbidity and mortality worldwide. Gastric varices occur in up to 30% of patients with cirrhosis, and they can rupture, leading to life-threatening bleeding. The clinical, epidemiological, and public health context of primary prophylaxis of gastric varices is therefore the need to prevent the development of this complication in patients at risk for cirrhosis and to reduce the associated morbidity and mortality. The clinical trials on primary prophylaxis of gastric varices are therefore focused on evaluating the safety and efficacy of various interventions, such as beta-blockers and endoscopic techniques, in reducing the risk of gastric varices in patients with cirrhosis. The goal of this trial is to find the most effective and safe strategies for primary prophylaxis of gastric varices, in order to improve the outcomes for patients with cirrhosis.

DETAILED DESCRIPTION:
Primary gastric varices (GV) are a condition that affects 17% of patients with liver cirrhosis who have not previously received treatment, either endoscopic or pharmacologic. Although the incidence of GV is lower than oesophageal varices (EV) and the bleeding rate is also less frequent, GV bleeding is more severe and is associated with higher re-bleeding and death rates when compared to EV. The management of acute GV bleeding is well established, but the primary prophylaxis (PP) for certain types of GV remains unclear. The management of GOV-1 (gastroesophageal varices type 1) is recommended as for EV, but for isolated gastric varices type 1 (IGV-1) and gastroesophageal varices type 2 (GOV-2), PP is not clearly defined. Existing guidelines from the American Association for the Study of Liver Diseases (AASLD) and the European Association for the Study of the Liver (EASL) do not provide strong recommendations for primary prophylaxis of IGV-1/GOV-2. While EASL suggests the use of nonselective beta-blockers (NSBB) for IGV-1/ GOV-2 based on one Randomized Controlled Trial (RCT) from 2011 on 89 patients, comparing NSBB vs. endoscopic glue injection for primary prophylaxis in GOV-2/IGV-1. The Baveno consensus VII recommends NSBB in PP but emphasizes the need for further studies. However, no study compares NSBB vs. EUS-GV management in primary prophylaxis. Establishing primary prophylaxis for IGV-1/GOV-2 is even more important as the 2-year incidence of variceal bleeding from IGV1 and GOV-2 type of varices is more frequent and profuse (78% and 54%, respectively) than the lesser curve (GOV-1) varices (28%).

Clinical research has shown that the use of non-selective beta-blockers, such as propranolol and nadolol, can be effective in reducing the risk of developing gastric varices in patients with cirrhosis. These medications work by reducing blood flow to the dilated veins in the stomach, thereby reducing the pressure in these vessels. In addition to the use of beta-blockers, there have been other interventions studied for primary prophylaxis of gastric varices. These include the use of endoscopic techniques such as band ligation and injection sclerotherapy, and the use of the cyanoacrylate glue.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Referred to St. Michael's Hospital (SMH) for esophagogastroduodenoscopy (EGD) screening for varices
* Patients with GOV-2 or IGV-1 varices with the size ≥ 10 mm

Exclusion Criteria:

* Age >75 and < 18 years
* Pregnancy
* Contraindications to beta-blockers and cyanoacrylate injection
* Prior treatment for prevention of bleeding from patients on beta-blockers
* Hepatic encephalopathy grade III/IV
* Hepatorenal syndrome, hepatocellular carcinoma, presence of deep jaundice (serum bilirubin >170 mmol/L)
* Cardiorespiratory failure
* Co-existing large oesophageal varices which require endoscopic intervention
* Child-Pugh C (score of 10-15 indicating decompensated disease)
* Presence of serious complications of liver cirrhosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of NSBB (Propanolol), EUS-guided combined therapy (coils + glue) of GOV-2 and IGV-1 | 3 months
  - incidence of bleeding during the follow-up
Assessment of NSBB (Propanolol), EUS-guided combined therapy (coils + glue) of GOV-2 and IGV-1 | 3 months
  -regression of gastric varices
Assessment of NSBB (Propanolol), EUS-guided combined therapy (coils + glue) of GOV-2 and IGV-1 | 6 months
  - incidence of bleeding during the follow-up
Assessment of NSBB (Propanolol), EUS-guided combined therapy (coils + glue) of GOV-2 and IGV-1 | 6 months
  -regression of gastric varices
Assessment of NSBB (Propanolol), EUS-guided combined therapy (coils + glue) of GOV-2 and IGV-1 | 9 months
  - incidence of bleeding during the follow-up
Assessment of NSBB (Propanolol), EUS-guided combined therapy (coils + glue) of GOV-2 and IGV-1 | 9 months
  -regression of gastric varices

SECONDARY OUTCOMES:
Estimation if any of the study arms is better for regression in size of varix | 3 months
  Assessing Size of Varix (mm)
Estimation if any of the study arms is better for regression in size of varix | 6 months
  Assessing Size of Varix (mm)
Estimation if any of the study arms is better for regression in size of varix | 9 months
  Assessing Size of Varix (mm)

OTHER OUTCOMES:
Safety of the procedure | - Follow-up visit after 3 months
  -Adverse Event (AE) rate for both methods
Safety of the procedure | - Follow-up visit after 6 months
  -AE rate for both methods
Safety of the procedure | - Follow-up visit after 9 months
  -AE rate for both methods

CONTACTS AND LOCATIONS:
Overall Officials: Samir C Grover, MD, MEd, Principal Investigator — Unity Health Toronto; Kareem Khalaf, HBSc, MD, Study Director — Unity Health Toronto; Nikko Gimpaya, HBSc, MEd, Study Director — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No